CLINICAL TRIAL: NCT03348800
Title: Anesthesia in Pediatric Dental Surgery: Effects of a Computer Controlled Delivery System on Pain and Heart Rate. A Randomized Clinical Trial
Brief Title: Evaluation of Pain Perception and Heart Rate in Children Who Received Dental Anesthesia
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Dr. Romeo Patini, DDS, PhD, Post Graduate Diploma in Oral Surgery, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP-01
Record Dates: First submitted 2017-11-13; First posted 2017-11-21 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Dental Anxiety
Keywords: Child; RCT; Anesthesia; Tooth extraction
MeSH Terms: interventions — Anesthesia, Dental

STUDY DESIGN:
Intervention Model Description: This study has a split-mouth model so participants will be anesthetized in one half of the maxilla with a conventional syringe and in the other half with the computer controlled delivery system.
  The anesthetic techniques will be the same in the two haves.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blindfolded during the tooth extractions and the outcome assessors will be unaware of dental procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Side (Experimental): The side in which computer controlled anesthetic delivery system will be used as dental anesthesia before dental surgery
  Interventions: Procedure: Dental anesthesia
- Control Side (Active Comparator): The side in which conventional syringe will be used as dental anesthesia before dental surgery
  Interventions: Procedure: Dental anesthesia

INTERVENTIONS:
Procedure: Dental anesthesia — A tooth extraction will be performed
  Other Names: Device: computer controlled delivery system named Wand®

SUMMARY:
The aim of this single-blind split-mouth study is to compare traditional syringe technique versus computer-controlled Wand® anesthetic System to evaluate pain perception, assessed with Visual Numerical Rating Scale, and heart rate in children requiring at least two tooth extractions on opposite sides of the maxilla. The investigators suppose that the feeling of fear during anesthesia administration is related to the use of the conventional syringe and that the pain to the lack of control of the plunger of the syringe.

The computer-controlled delivery system allows the operator to hide the needle and to control the pressure exerted during anesthetic administration.

DETAILED DESCRIPTION:
The sample of this single-blind split mouth study will be made up of 76 consecutive children (38 men and 38 female) between 5 and 12 years attending the Paediatric Dentistry Unit of Catholic University of Sacred Heart, Rome, Italy, from November 2016 for routinary dental treatments who needed at least two dental extractions on both left and right maxillary arches. The participants will have to be in good general health state with no contraindications to local anesthetics. Exclusion criteria are: suffering from any medical condition that could alter pain perception or taking any antibiotic or antinflammatory drugs in the last month before the procedures. A detailed informed written consent form will be signed by each patient's parent or guardian of children enrolled in this study before every clinical procedure. Patients will be informed that a computer controlled and traditional syringe techniques will be used for their dental procedures. No patients should have previously experienced a conventional syringe technique nor the Wand® injection. The sample size was calculated performing a power analysis based on the results of previous studies to detect at least a 1 grade Numerical Visual Rating Scale difference with Standard Deviation of 1.05 and at least a 3 mmHg difference with Standard Deviation of 4 mmHg between groups. The alpha and beta values were set as 0.01 and 0.95 respectively and the sample size was calculated to be 30 subjects for each group.

MEASURES Pain perception will be explained to patients before injections. The Numerical Visual Rating Scale is a pain scale based on Visual rating scale and Numerical rating scale that was used for the same purpose on adults in a previous report. This scale demonstrated to be easier to understand by the patients and was preferred to other scales that could have caused difficulties in evaluation by the children. Heart rate will be assessed using a pulse oximeter before and after the injection.

PROCEDURES One half of the maxilla will be anesthetized using the Wand® system and the contralateral half by a conventional syringe. In both halves the intraligamentary technique will be the sole used. Anesthesia will be administered by the same previously calibrated operator. The order of techniques will be randomly selected. Randomization will be obtained through a random sequence generated by a Personal Computer. A distraction technique for palatal injections, in the form of pressure applied using the handle of the dental mirror, will be used before needle's insertion in both techniques. Following the intraligamentary technique the needle will be inserted parallel to the long axis of the tooth into the sulcus of each root and some drops of the local anesthetic solution will be administered before the needle entered the tissue. After few seconds the needle will be advanced penetrating the tissue and an additional amount of solution will be administered. The Wand® will be set on a pre-programmed injection mode named "Single Tooth Anesthesia" (speed mode 0,005 mL/sec). Once anesthesia will be achieved, tooth extractions will be performed. Patients should have been previously blindfolded with a commonly used sleeping mask so they will not distinguish which anesthetic delivery system was being used. Anesthesia procedures and tooth extractions will be completed in the same session according to a split-mouth design. The Wand® system produces audible beeps that will be deactivated. Immediately after delivery of local anesthetic, children will be asked to remove their mask and rate the pain felt during the anesthetic administration.

All patients will receive mepivacaine 3% with a vasoconstrictor (Carbocaine 20 mg/ml with epinephrine 1:100.000 Dentsply Italy srl). A 1.8 mL anesthetic cartridge will be used for both procedures (Wand® vs. traditional). The local anesthetic will be injected with an extra-short 30 gauge dental needle for both Wand® (30 G handpiece and needle, Milestone Scientific) and with a traditional 30 Gauge needle (Trend Ject 0.30x21mm) for conventional injections.

The following data will be collected through the use of a structured form:

1. Patient's age
2. Patient's gender
3. Number of tooth/teeth extracted
4. Score on Visual numerical Rating Scale
5. Heart Rate before injection
6. Heart Rate after injection

STATISTICAL ANALYSIS All analyses will be performed using a commercially available software program (SPSS®, version 20.0, SPSS Inc., Chicago, Illinois, USA). Exploratory statistics revealed that all variables were normally distributed with equality of variances.

Pain perception and Heart Rate changes during injection will be evaluated and paired t-test will be used to assess statistical significance for each outcome. All comparisons will be considered significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* good general health state and no contraindications to local anesthetics

Exclusion Criteria:

* suffering from any medical condition that could alter pain perception or taking any antibiotic or antinflammatory drugs in the last month before the procedures

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Pain felt during dental anesthesia | 2 minutes after dental anesthesia
  Pain will be assessed with the use of a (VNRS) Visual Numerical Rating Scale. Such Scale ranges from 0 to 10 with 0 meaning "no pain" and 10 meaning "the worst pain possible".

SECONDARY OUTCOMES:
Heart Rate during dental anesthesia | 2 minutes after and 2 minutes before dental anesthesia
  Heart Rate will be assessed with the use of a pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Cordaro, MD, Dean, Study Chair — Catholic University of Sacred Heart
Locations (1):
- Catholic University of Sacred Heart, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garret-Bernardin A, Cantile T, D'Anto V, Galanakis A, Fauxpoint G, Ferrazzano GF, De Rosa S, Vallogini G, Romeo U, Galeotti A. Pain Experience and Behavior Management in Pediatric Dentistry: A Comparison between Traditional Local Anesthesia and the Wand Computerized Delivery System. Pain Res Manag. 2017;2017:7941238. doi: 10.1155/2017/7941238. Epub 2017 Feb 15. PMID 28293129
- [Result] Patini R, Coviello V, Raffaelli L, Manicone PF, Dehkhargani SZ, Verdugo F, Perfetti G, D'Addona A. Subjective pain response to two anesthetic systems in dental surgery: traditional syringe vs. a computer controlled delivery system. J Biol Regul Homeost Agents. 2012 Apr-Jun;26(2 Suppl):89-97. PMID 23164333